CLINICAL TRIAL: NCT04839653
Title: Efficacy and Safety of Selective Digestive Decontamination in the ICU With Rates of Antibiotic-resistant Bacteria
Brief Title: Efficacy and Safety of Selective Digestive Decontamination in the ICU With High Rates of Antibiotic-resistant Bacteria
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MEDSI Clinical Hospital 1, ICU (Other)
Responsible Party: Principal Investigator, Yury Surovoy, Principal Investigator, MEDSI Clinical Hospital 1, ICU
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SDDMEDSI2021
Record Dates: First submitted 2021-04-05; First posted 2021-04-09 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Pneumonia, Ventilator-Associated; Pneumonia; Bloodstream Infection; Sepsis; Respiratory Distress Syndrome; Respiratory Tract Infections; Critical Illness
Keywords: Pneumonia; Ventilator-Associated Pneumonia; Selective Digestive Decontamination; Secondary Infections; Infection prophylaxis; Bloodstream Infection
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Pneumonia; Sepsis; Respiratory Distress Syndrome; Respiratory Tract Infections; Critical Illness; Coinfection | interventions — Polymyxin B; Gentamicins; Suspensions; Vancomycin; Ceftriaxone; Cefotaxime

STUDY DESIGN:
Intervention Model Description: During the first period patients will receive standard care. During the second period SDD protocol will be implemented.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group: standard care (No Intervention): Patients in the standard care group will be prospectively evaluated to determine pre-defined clinical outcomes.
- Selective digestive decontamination group (Experimental): 1. Oral paste (0,5 g) containing 10 mg of polymyxin B, 10 mg of gentamycin and 150 mg of amphotericine B q6h
  2. In the NGT 10 ml of suspension containing 100 mg of polymyxin B, 80 mg of gentamycin, 350 mg of amphotericine B and 500 mg of vancomycin q6h
  3. A 3-day course of intravenous cefotaxime 1 g q6h/ceftriaxone 1 qd
  Interventions: Drug: Oral Paste(0,5 g) containing 10 mg of polymyxin B, 10 mg of gentamycin and 150 mg of amphotericine B or 500 000 U of nistatin q6h; Drug: Suspension (10 ml) containing 100 mg of polymyxin B, 80 mg of gentamycin, 350 mg of amphotericine B or 8000000 U of nistation and 500 mg of vancomycin q6h; Drug: Intravenous Antibacterial Agent - a 3-day course of systemic cefotaxime 1 g q6h or ceftriaxone 1 g qd

INTERVENTIONS:
Drug: Oral Paste(0,5 g) containing 10 mg of polymyxin B, 10 mg of gentamycin and 150 mg of amphotericine B or 500 000 U of nistatin q6h — The oral paste will be applied topically on the oropharyngeal mucosa q6h.
  Other Names: Polymyxin B, Gentamycin, Amphotericine B, Nistatin
  Arms: Selective digestive decontamination group
Drug: Suspension (10 ml) containing 100 mg of polymyxin B, 80 mg of gentamycin, 350 mg of amphotericine B or 8000000 U of nistation and 500 mg of vancomycin q6h — The suspension will be administered through the nasogastric tube q6h.
  Other Names: Polymyxin B, Gentamycin, Amphotericine B, Vancomycine, Nistatin
  Arms: Selective digestive decontamination group
Drug: Intravenous Antibacterial Agent - a 3-day course of systemic cefotaxime 1 g q6h or ceftriaxone 1 g qd — Patients who do not receive systemic antibiotics for other reasons will get a short course of systemic antibiotic
  Other Names: Cefotaxime, Ceftriaxone
  Arms: Selective digestive decontamination group

SUMMARY:
Secondary infections remain a major cause of mortality in critically ill patients, mainly because of high prevalence of multidrug-resistant microorganisms. Therefore strategies aimed to reduce the incidence of ventilator-associated pneumoniae (VAP) and bloodstream infections are of utmost important. There is robust data on selective digestive decontamination (SDD) efficacy in reduction of secondary infections in intensive care units (ICU) with low rates of antibacterial resistance. However the data received from hospitals with moderate-to-high rates of resistance is equivocal.

This as an interventional parallel open-label study investigating the effect of selective digestive decontamination on the rates of ventilator-associated pneumonia in critically ill patients admitted to the ICU with high prevalence of drug-resistant bacteria. Secondary outcomes include rates of bloodstream infections, mortality, duration of mechanical ventilation, duration of ICU stay, resistance selection and overall antibiotic consumption.

DETAILED DESCRIPTION:
Single-center prospective interventional parallel study. During the first period of the study patients will receive standard therapy. During the second period the SDD protocol will be implemented in addition to the standard care. The first period will end at the moment of the last admitted patient ICU discharge or death.

Study population: general ICU adult patients anticipated to receive prolonged mechanical ventilation (more than 48 hours). Patients who are terminally ill and are anticipated to die in the next 24 hours will be excluded, so are patients with malignancies (except for patients with primary central nervous system tumors who received radical treatment) and patients admitted from other hospitals who received mechanical ventilation (including non-invasive ventilation) for more than 24 hours.

Patients in the interventional arm will receive the following SDD protocol:

1. Oral paste (0,5 g) containing 10 mg of polymyxin B, 10 mg of gentamycin and 150 mg of amphotericine B/500000 U of nistatin q6h
2. In the nasogastric tube (NGT) 10 ml of suspension containing 100 mg of polymyxin B, 80 mg of gentamycin, 350 mg of amphotericine B/8000000 U of nistatin and 500 mg of vancomycin q6h
3. A 3-day course of intravenous cefotaxime 1 g q6h/ceftriaxone 1 qd

Statistical considerations and recruitment plant: VAP incidence in the ICU with high rates of antibacterial resistance is 16,7 event per 1000 days of MV. To reveal a 25% decrease of VAP events (power 80%, p < 0,05) the study should recruit 25 patients in each group. However because of the poor prognosis in mechanically ventilated elderly patients especially in the setting of acute respiratory distress syndrome the goal is to recruit in each arm at least 25 patients younger than 65 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with expected MV for more than 24 hours

Exclusion Criteria:

* Moribund condition and expected death within 24 hours
* Malignancy (excluding primary CNS tumors)
* Patients transferred from other hospitals who were mechanically ventilated for more than 24 hours (including NIV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
The incidence of ventilator-associated pneumonia | During ICU stay up to 28 days
  Number of ventilator-associated pneumonia events per 1000 days of MV

SECONDARY OUTCOMES:
The incidence of bloodstream infections | During ICU stay up to 28 days
  Number of bloodstream infection events per 1000 days of ICU stay
ICU mortality | During ICU stay up to 28 days
  All-cause mortality
Duration of mechanical ventilation | During ICU stay up to 28 days
  The duration that the patient receives mechanical ventilation in the ICU
Duration of organ support | During ICU stay up to 28 days
  The duration that the patient receives mechanical ventilation, vasopressor infusion or renal-replacement therapy
Antimicrobial drug consumption | During ICU stay up to 28 days
  Average antimicrobial drug consumption (as daily defined doses) per patient stay
Antimicrobial resistance selection | During ICU stay up to 28 days
  The magnitude of antimicrobial resistance selection in terms of resistant microorganisms prevalence and whole burden of AMR genes

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Azovskiy, MD, phD, Principal Investigator — MEDSI Clinical Hospital 1
Locations (1):
- MEDSI Clinical Hospital 1, Moscow, Russia